CLINICAL TRIAL: NCT04919226
Title: A Prospective, Randomised, Controlled, Open-label, Multicentre Study to Evaluate Efficacy, Safety and Patient-Reported Outcomes of Peptide Receptor Radionuclide Therapy (PRRT) With 177Lu-Edotreotide Compared to Best Standard of Care in Patients With Well-differentiated Aggressive Grade 2 and Grade 3, Somatostatin Receptor-Positive (SSTR+), Neuroendocrine Tumours of GastroEnteric or Pancreatic Origin
Brief Title: Lutetium 177Lu-Edotreotide Versus Best Standard of Care in Well-differentiated Aggressive Grade-2 and Grade-3 GastroEnteroPancreatic NeuroEndocrine Tumors (GEP-NETs) - COMPOSE
Acronym: COMPOSE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ITM Solucin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP-1111-02CT
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumors
Keywords: GastroEnteroPancreatic; non-functional and functional GastroEnteroPancreatic NeuroEndocrine Tumors (GEP-NET)
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-; Capecitabine; Temozolomide; amino-acid, glucose, and electrolyte solution; Everolimus; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peptide Receptor Radionuclide Therapy (PRRT) Arm (Experimental)
  Interventions: Drug: 177Lu-Edotreotide (Peptide Receptor Radionuclide Therapy) PRRT; Other: Amino-Acid Solution
- CAPTEM(Capecitabine-Temozolomide), Everolimus, FOLFOX(Folinic acid + Fluorouracil + Oxaliplatin) (Active Comparator)
  Interventions: Drug: CAPTEM (Capecitabine and Temozolomide); Drug: Everolimus; Drug: FOLFOX (Folinic acid + Fluorouracil + Oxaliplatin)

INTERVENTIONS:
Drug: 177Lu-Edotreotide (Peptide Receptor Radionuclide Therapy) PRRT — Peptide Receptor Radionuclide Therapy (PRRT) using 177Lu-edotreotide with a defined number of cycles will be administered.
  Other Names: 177Lu-DOTATOC 177Lu-Edo
  Arms: Peptide Receptor Radionuclide Therapy (PRRT) Arm
Drug: CAPTEM (Capecitabine and Temozolomide) — Best standard of care treatment (investigator's choice [from the protocol comparator list]) according to individual risk-benefit assessment, institutional protocols, the local Prescribing Information, local regulations, or the local guidelines.
  Arms: CAPTEM(Capecitabine-Temozolomide), Everolimus, FOLFOX(Folinic acid + Fluorouracil + Oxaliplatin)
Other: Amino-Acid Solution — The Amino-Acid Solution (AAS) to be used in this study will contain a mixture of lysine and arginine diluted in an electrolyte solution.
  Other Names: Arginine-Lysine Solution
  Arms: Peptide Receptor Radionuclide Therapy (PRRT) Arm
Drug: Everolimus — Best standard of care treatment (investigator's choice [from the protocol comparator list]) according to individual risk-benefit assessment, institutional protocols, the local Prescribing Information, local regulations, or the local guidelines.
  Arms: CAPTEM(Capecitabine-Temozolomide), Everolimus, FOLFOX(Folinic acid + Fluorouracil + Oxaliplatin)
Drug: FOLFOX (Folinic acid + Fluorouracil + Oxaliplatin) — Best standard of care treatment (investigator's choice [from the protocol comparator list]) according to individual risk-benefit assessment, institutional protocols, the local Prescribing Information, local regulations, or the local guidelines.
  Arms: CAPTEM(Capecitabine-Temozolomide), Everolimus, FOLFOX(Folinic acid + Fluorouracil + Oxaliplatin)

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety & patient-reported outcomes of peptide receptor radionuclide therapy (PRRT) with 177Lu-Edotreotide as 1st or 2nd line of treatment compared to best standard of care in patients with well-differentiated aggressive grade 2 and grade 3, somatostatin receptor-positive (SSTR+), neuroendocrine tumours of gastroenteric or pancreatic origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Histologically confirmed diagnosis of unresectable, well-differentiated GastroEnteroPancreatic NeuroEndocrine Tumors (GEP-NETs). measurable site of disease per RECIST v1.1 (Response evaluation criteria in solid tumors) using contrast computed tomography (CT) / magnetic resonance imaging (MRI).
* Somatostatin receptor-positive (SSTR+) disease.

Exclusion Criteria:

* Known hypersensitivity to Lutetium 177Lu, edotreotide, DOTA (dodecane tetraacetic acid), any of the comparators, or any excipient or derivative (e.g. rapamycin).
* Prior (Peptide Receptor Radionuclide Therapy) PRRT.
* Any major surgery within 4 weeks prior to randomization in the trial.
* Therapy with an investigational compound and/or medical device within 30 days or 7 half-life periods (whichever is longer) prior to randomization.
* Other known malignancies.
* Serious non-malignant disease.
* Renal, hepatic, cardiovascular, or hematological organ dysfunction, potentially interfering with the safety of the trial treatments.
* Pregnant or breastfeeding women.
* Patients not able to declare meaningful informed consent on their own or any other vulnerable population to that.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Every 12 weeks from randomization until disease progression or death whichever occurs earlier, during the time necessary to observe 148 Progression Free Survival (PFS) events.
  PFS (Progression-Free Survival), defined as the time from randomization until documented RECIST v1.1 (Response evaluation criteria in solid tumors) progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | Up to 3 years after disease progression, or to a maximum of 5 years after randomization
  OS (Overall Survival), defined as the time from randomization until death;

CONTACTS AND LOCATIONS:
Locations (42):
- United States (14):
  - Stanford Cancer Center, Palo Alto, California
  - University of Colorado Hospital, Nuclear Medicine, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Department of Oncology, Rochester, Minnesota
  - Washington University Alvin J. Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - ICAHN School of Medicine at Mount Sinai, Tish Cancer Institute, New York, New York
  - Duke University School of Medicine, Duke Cancer Institute, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai
  - Affiliated Hospital of Jiangnan University, Wuxi
- France (4):
  - Haut-Leveque Hospital, Department of Hepatogastroenterology and Digestive Tract Oncology, Pessac, Bordeaux
  - Nantes University Hospital Center - Hotel Dieu Hospital, Nantes, Cedex
  - Edouard Herriot Hospital, Medical Oncology Unit, Lyon
  - IUCT Oncopole - Institut Universitaire du Cancer de Toulouse, Toulouse
- Germany (4):
  - Charite - University Hospital Berlin, Berlin
  - University Hospital Bonn, Department of Nuclear Medicine, Bonn
  - University Hospital Erlangen, Department of Internal Medicine I - Endocrinology, Erlangen
  - University Duisburg-Essen, University Hospital Essen, Clinic for Nuclear Medicine, Essen
- India (3):
  - HCG Cancer Centre, Medical Oncology, Bangalore, Karnataka
  - All India Institute Of Medical Sciences, Nuclear Medicine, New Delhi, National Capital Territory of Delhi
  - Tata Memorial Hospital, Nuclear Medicine & Molecular Imaging, Mumbai
- Italy (3):
  - University Polyclinic Hospital "G. Martino", Department of Biomedical Sciences, Dentistry and Morphological and Functional Imaging, Complex Operational Unit of Nuclear Medicine, Messina
  - European Institute of Oncology (IEO), IRCCS, Milan
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Complex Operative Unit of Medical Oncology, Rome
- Netherlands (2):
  - VU Medical Center (VUMC), Department of Medical Oncology, Amsterdam
  - Erasmus University Medical Center Rotterdam, Rotterdam
- Spain (7):
  - University Hospital Vall d'Hebron, Department of Medical Oncology, Barcelona
  - ICO Hospitalet, Catalan Institute of Oncology, Barcelona
  - University General Hospital Gregorio Maranon, Madrid
  - University Hospital 12 de Octubre, Department of Gastroenterology, Madrid
  - Central University Hospital de Asturias (HUCA), IUOPA - Universitary Institute of Oncology, Oviedo
  - University Hospital Complex of Santiago (CHUS), Santiago de Compostela
  - University and Polytechnic Hospital La Fe, Endocrinology, Valencia
- King's College Hospital, London, United Kingdom